CLINICAL TRIAL: NCT01936246
Title: Protein Supplementation in Infants With Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CCHMCProtein
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Perinatal Stroke; Hypoxic-ischemic Encephalopathy; White Matter Injury
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Increased protein (Experimental): Full term infants will be on 4 g/kg/day of protein. Preterm infants will be on 4.5 g/kg/day of protein until term corrected age. Beneprotein powder will be used; if this is not tolerated, Complete Amino Acids will be used. Max protein will be 30 g/day. Increased protein will be given until 12 months corrected age.
  Interventions: Dietary Supplement: Increased protein
- Standard diet (No Intervention): Infants will be given a usual diet. If infants in this arm have poor growth, protein or caloric supplementation may be given per the discretion of the clinical team.

INTERVENTIONS:
Dietary Supplement: Increased protein
  Other Names: Beneprotein or Complete Amino Acids
  Arms: Increased protein

SUMMARY:
To date, few studies have been done regarding nutrition supplementation in infants with brain injury. Therefore, the investigators are proposing to study the effects of protein supplementation in this group of babies. The investigators will recruit 24 infants with brain injury (evidence of hemorrhage, white matter injury, or gray matter injury) admitted to the Cincinnati Children's Hospital Neonatal Intensive Care Unit (NICU) into the study. Upon diagnosis, the investigators will obtain consent from the parents for participation in the study, then randomly assign the baby to one of two groups - an increased protein group and a control group. Both groups of infants will be monitored to ensure no adverse effects occur due to the supplementation.

Protein supplementation will continue for the first 12 months of age. Growth parameters, such as weight, length, and head circumference, will be measured while the infant is the NICU. Head circumference will be measured in the investigators outpatient clinic at three, six, and 12 months of age. At 18-22 months, the infants will be tested for neurodevelopmental outcomes using the Bayley Scales of Infant Development. The investigators hypothesize that infants who receive the additional protein will demonstrate increased head growth and improved neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the NICU at CCHMC
* Known or suspected brain injury
* Parental consent obtained
* At least 48 hours of age at the time of randomization

Exclusion Criteria:

* Congenital or posthemorrhagic hydrocephalus
* Major congenital brain malformations
* Congenital gastrointestinal malformations or Bell Stage III NEC
* Inborn errors of metabolism
* Chromosomal abnormalities
* Significant cardiac disease

Ages: 2 Days to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Head circumference | 12 months of age +/- 4 weeks

SECONDARY OUTCOMES:
Neurodevelopmental outcome on Bayley Scales of Infant Development | 18-22 months
Weight and length | 3, 6, 12 months of age

OTHER OUTCOMES:
Blood urea nitrogen | 10 and 30 days post study initiation
CO2 from renal panel | 10 and 30 days post study initiation
  To assess for metabolic acidosis

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Merhar, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Merhar SL, Meinzen-Derr J, Sprague J, Wessel JJ, Leugers S, Painter J, Valentine CJ. Safety and Tolerability of Enteral Protein Supplementation for Infants With Brain Injury. Nutr Clin Pract. 2015 Aug;30(4):546-50. doi: 10.1177/0884533614567715. Epub 2015 Jan 23. PMID 25616519